CLINICAL TRIAL: NCT06895434
Title: Does Balneotherapy Affect Blood Pressure and Pulse?
Brief Title: Effect of Repeated Thermomineral Water Immersion on Blood Pressure and Heart Rate in Individuals with Chronic Pain Due to Musculoskeletal System Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Collaborators: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Balneotherapy +Blood Pressure
Record Dates: First submitted 2024-02-05; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-02

CONDITIONS: Balneology; Blood Pressure; Heart Rate
Keywords: Balneotherapy; Blood Pressure; Cardiac Rate
MeSH Terms: interventions — Balneology; Physical Therapy Modalities; Transcutaneous Electric Nerve Stimulation; Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Balneotherapy with physical therapy (Active Comparator): Balneotherapy applied in the thermal pools to patients for 20 minutes, at a temperature of 38-40°C. After resting for 30 minutes,physical therapy was applied.
  Interventions: Other: Balneotherapy with physical therapy
- Only physical therapy (Active Comparator): Patients in group 2 were applied only a physical therapy program.
  Interventions: Other: Physical therapy

INTERVENTIONS:
Other: Balneotherapy with physical therapy — Balneotherapy applied in the thermal pools to patients for 20 minutes, at a temperature of 38-40°C. After resting for 30 minutes,physical therapy was applied.
  A physical therapy program (5 days a week for 2 weeks, a total of 10 sessions) was applied to the painful area, including 20 minutes of hot pack at 60°C, 20 minutes of conventional TENS at 80 Hz and US at 3 MHz frequency and 1.5 watt/cm2 intensity.
  Other Names: Transcutaneous Electrical Nerve Stimulation (TENS); Hot Pack; Ultrasound(US) Therapy
  Arms: Balneotherapy with physical therapy
Other: Physical therapy — A physical therapy program (5 days a week for 2 weeks, a total of 10 sessions) was applied to the painful area, including 20 minutes of hot pack at 60°C, 20 minutes of conventional TENS at 80 Hz and US at 3 MHz frequency and 1.5 watt/cm2 intensity.
  Other Names: Transcutaneous Electrical Nerve Stimulation (TENS); Hot Pack; Ultrasound(US) Therapy
  Arms: Only physical therapy

SUMMARY:
Purpose: This study aimed to investigate the effect of balneotherapy on blood pressure and heart rate in patients.

Methods: A total of 240 participants who met the inclusion criteria of the study were divided into 2 groups (120 participants in each group).

A 10-session physical therapy was applied to all participants in both groups. Balneotherapy was applied to Group I.

The participants filled out a questionnaire containing demographic data, and participants arterial blood pressures and heart rate were measured and recorded before and after treatment throughout the treatment.

DETAILED DESCRIPTION:
INTRODUCTION: Spa treatment is an additional and auxiliary method that has an important place in the prevention, treatment and rehabilitation of a wide variety of diseases. The majority of people who go to thermal springs for treatment have rheumatic diseases, followed by dermatological, gastrointestinal and gynecological diseases. However, outside these disease groups, the place of spa treatment and its most basic element, thermomineral water and mud, that is, balneotherapy, is increasing.

Answers to questions such as in what direction and how these factors affect a human organism in water (during immersion) form the basis of balneotherapy in cardiovascular diseases. For this purpose, the investigators planned to investigate the effects of balneotherapy on blood pressure and heart rate in patients.

METHODS The study was designed as a prospective, randomized, controlled, and single-blind study. A total of 240 participants who applied to the medical ecology and hydroclimatology and physical therapy and rehabilitation outpatient clinic with pain complaints, met the study criteria and signed the participants information consent form were included in the study.

A total of 240 participants who met the inclusion criteria of the study were divided into 2 groups (120 participants in each group) with simple randomization method by using a table of random numbers created on the computer. The researchers who made the assessment measurements were unaware of which participant was in which group. Statistical analysis of the results was performed by a biostatistician who had no information about the therapies the participant groups received.

All participants in both groups underwent a 10-session physical therapy program (e.g. Hot pack, TENS, ultrasound, etc.) to the areas of pain. Balneotherapy was applied to group I before treatment. Balneotherapy applied in the thermal pools to patients for 20 minutes, at a temperature of 38-40°C. After resting for 30 minutes,physical therapy was applied.

The participants filled out a questionnaire containing demographic data, and arterial blood pressures and heart rate were measured and recorded before and after treatment throughout the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 45 and 75
* Patients with pain associated with rheumatic diseases

Exclusion Criteria:

* Inflammatory rheumatic disease (rheumatoid arthritis, ankylosing spondylitis, etc.),
* Diagnosed with uncontrolled arterial hypertension and diabetes mellitus,
* Having a diagnosed neuro-psychiatric problem,
* Undergoing malignancy treatment,
* Having a bleeding disease,
* Having an infectious disease with fever,
* Patients who received physical therapy, balneotherapy or both in the last six mounths.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Blood pressure and heart rate | Measurements were made on the individuals included in the study from the beginning to the end of the treatment protocol (on the days of treatment - 10 days in total).
  Only blood pressure and heart rate measurements were made of the participants, no other measurements or evaluations were made. Blood pressure and heart rate were measured in all patients before starting their treatment and at the end of the treatment, after 30 minutes of rest.
  Blood pressure and heart rate was evaluated with a non invasive sphygmomanometer on the same arm (right) (OMRON HBP-1320).
  The pulse number was confirmed by measuring with the researcher's three fingers on the radial artery.

CONTACTS AND LOCATIONS:
Overall Officials: Kağan Özkuk, Study Director — Uşak University
Locations (1):
- UsakU, Merkez, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No